CLINICAL TRIAL: NCT02670746
Title: Non-interventional Observational Post-authorization Study to Assess Clinical and Patient Reported Outcomes With Nab-paclitaxel in Combination With Gemcitabine in Routine Clinical Practice Treating Pancreatic Cancer (TRUST)
Brief Title: A Study to Assess Clinical an Patient Reported Outcomes With Nab-paclitaxel in Combination With Gemcitabine in Route Clinical Practice Treating Pancreatic Cancer
Acronym: TRUST
Status: Terminated | Type: Observational
Why Stopped: Due to slow recruitment study is being terminated.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: ABI-007-PANC-008
Record Dates: First submitted 2015-08-31; First posted 2016-02-02 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic Cancer; Observational; Nab-Paclitaxel; Abraxane; ABI-007; Gemcitabine; Non-interventional; Netherlands; Quality of Life
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nab-paclitaxel in combination with gemcitabine (AG): The objective is to prospectively assess the use and treatment outcomes of nab-paclitaxel plus gemcitabine in pancreatic ductal adenocarcinoma. In all cases, the decision to treat the patient with nab-paclitaxel in combination with gemcitabine was already made prior to the decision to enter the subject into the study. Treatment will be according to routine clinical practice and based on recommendations as per Summary of Product Characteristics (SPC).

SUMMARY:
The objective of the study is to prospectively assess the use and treatment outcomes of nab-paclitaxel plus gemcitabine in pancreatic ductal adenocarcinoma in the Netherlands. Additional objectives are to monitor the incidence and reversibility of neuropathy during treatment, to assess the patient's Quality of life when treated with nab-paclitaxel/gemcitabine and to evaluate the use of resources that come with treating metastatic pancreatic cancer.

DETAILED DESCRIPTION:
The TRUST, a prospective, non-interventional observational single arm study with Nab-paclitaxel + Gemcitabine (NG) in pancreas carcinoma in the Netherlands, was started in 2015 to observe and register the daily use of Nab-paclitaxel. The primary objective was to prospectively assess safety of NG in metastatic pancreatic cancer under routine clinical practice. One of the major secondary objectives was to assess the influence of treatment with Nab-paclitaxel + Gemcitabine on the quality of life. The goal was to include 200 patients within a period of two year and collect their prospective data.

The study has included 44 patients in the period between October 2015 and October 2017. Of these patients, 41% were diagnosed with metastasized disease. 54% was diagnosed with local disease of which 18% was resectable and 36% was locally advanced. 73% of the patients with metastasized disease were treated with NG.

Over 70% of all NG treated patients received this treatment as a fist line of care. 21% of these patients had locally advanced pancreatic cancer. 20% of the patients had had a previous systemic treatment. Of all NG treated patients, 66% had an ECOG performance status of 0 or 1 and 62% of the patients was 75 years or younger.

At the time the study was terminated, 6 out of the 44 patients were still treated. 14 patients had stopped treatment due to disease progression, 8 patients had stopped due to adverse events and 7 patients had chosen to stop treatment.

The low inclusion rate, which led to a prospective study duration of 10 years, and the heterogenicity of the study population have led to the decision to terminate the study. Therefore, no analysis, apart from the detailed description of the study population above, can be performed.

All patients involved have taken the time to participate in the study and have filled out questionnaires. We would like to express our gratitude towards these patients.

We remain convinced that quality of life is an important parameter in pancreatic cancer which should be taken into consideration in daily care of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who understand and voluntarily sign an informed consent form.
* Patients treated for pancreatic adenocarcinoma.

Exclusion Criteria:

* Patients currently treated for metastatic pancreatic cancer with other therapy than nab-paclitaxel plus gemcitabine
* Refusal to participate in the study.
* Women who are pregnant or breast-feeding.
* Hypersensitivity to the active substance or to any of the excipients.
* Participation in interventional trials during the period of treatment with nab-paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two-hundred adult patients treated with the combination nab-paclitaxel and gemcitabine (AG) for metastatic pancreatic adenocarcinoma will be recruited from approximately 25 oncology sites in the Netherlands. In all cases, the decision to treat the patient with AG was already made prior to the decision to enter the subject into the study. Treatment will be according to routine clinical practice and based on recommendations as per SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to approximately 3 years
  Survival is defined as the time from the first dose of nab-paclitaxel in combination with gemcitabine date to the date of death (any cause).
Adverse Event (AE) | Up to approximately 3 years
  Adverse events will be classified using the MedDRA classification system. The severity of the toxicities will be graded according to the NCI CTCAE VERSION 4.03 whenever possible.

SECONDARY OUTCOMES:
Change from baseline in the EORTC-QLQ-CIPN-20 (European Organization for Research and Treatment of Cancer Quality of Life Instrument In Patients With Chemotherapy Induced Peripheral Neuropathy ) | up to approximately 3 years
  The instrument contains 20 questions evaluating sensory, motor, and autonomic symptoms, and has been validated as an assessment tool for CIPN. All scale scores are linearly converted to a 0-100 scale, with higher scores indicating more symptom burden.
Change from baseline in the EORTC-QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Instrument) | up to approximately 3 years
  The instrument contains 30 questions evaluating quality of life in cancer patients.
Change from baseline in the EuroQuality of Life : EQ5D-3L | up to approximately 3 years
  A generic Quality of Life (QOL) instrument to measure and evaluate health status outcomes. The 3 Level (3L) version describes general health based on five distinct dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 Levels (indicating no problem, some or moderate problem and extreme problem).
Evaluate the incidence of neuropathy - grade 1-5 | up to approximately 3 years
  Descriptive analysis of incidence and severity of neuropathy according to physicians assessment
Evaluate reversibility of neuropathy to Gr ≤1 | up to approximately 3 years
  The time to decrease of neuropathy to Gr ≤1 using the NCI CTCAE grading scale.
Evaluate the resources utilized for treatment of pancreatic adenocarcinoma with the combination nab-paclitaxel/gemcitabine in routine clinical practice | up to approximately 3 years
  Per hospital, one generalized questionnaire will be filled in to evaluate the use of utilized resources when treating metastatic pancreatic cancer within routine clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Stevens, Msc, Study Director — Celgene Corporation
Locations (18):
- Netherlands (18):
  - Rijnstate Ziekenhuis, Arnhem, Gelderland
  - Amphia ziekenhuis, Breda, Gelderland
  - Gelderse Vallei, Ede, North Brabant
  - Elkerliek Ziekenhuis, Helmond, North Brabant
  - Maxima Medisch Centrum, Veldhoven, North Brabant
  - BovenIJ Ziekenhuis, Amsterdam, North Holland
  - Academic Medical Centre, Amsterdam, North Holland
  - Spaarne Gasthuis, Haarlem, North Holland
  - Tergooi, Hilversum, North Holland
  - Isala, Zwolle, Overijssel
  - Ziekenhuis de Tjongerschans, Heerenveen, Provincie Friesland
  - Antonius Ziekenhuis Sneek, Sneek, Provincie Friesland
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - LUMC, Leiden, South Holland
  - HagaZiekenhuis, The Hague, South Holland
  - Zorgsaam Zeeuws -Vlaanderen, Terneuzen, Zeeland
  - Martini Ziekenhuis, Groningen
  - UMC Utrecht, Utrecht

REFERENCES:
- [Background] Reni M, Zanon S, Balzano G, Passoni P, Pircher C, Chiaravalli M, Fugazza C, Ceraulo D, Nicoletti R, Arcidiacono PG, Macchini M, Peretti U, Castoldi R, Doglioni C, Falconi M, Partelli S, Gianni L. A randomised phase 2 trial of nab-paclitaxel plus gemcitabine with or without capecitabine and cisplatin in locally advanced or borderline resectable pancreatic adenocarcinoma. Eur J Cancer. 2018 Oct;102:95-102. doi: 10.1016/j.ejca.2018.07.007. Epub 2018 Aug 24. PMID 30149366
- [Background] Vogl DT, Raje N, Jagannath S, Richardson P, Hari P, Orlowski R, Supko JG, Tamang D, Yang M, Jones SS, Wheeler C, Markelewicz RJ, Lonial S. Ricolinostat, the First Selective Histone Deacetylase 6 Inhibitor, in Combination with Bortezomib and Dexamethasone for Relapsed or Refractory Multiple Myeloma. Clin Cancer Res. 2017 Jul 1;23(13):3307-3315. doi: 10.1158/1078-0432.CCR-16-2526. Epub 2017 Jan 4. PMID 28053023
- [Background] Kim S, Signorovitch JE, Yang H, Patterson-Lomba O, Xiang CQ, Ung B, Parisi M, Marshall JL. Comparative Effectiveness of nab-Paclitaxel Plus Gemcitabine vs FOLFIRINOX in Metastatic Pancreatic Cancer: A Retrospective Nationwide Chart Review in the United States. Adv Ther. 2018 Oct;35(10):1564-1577. doi: 10.1007/s12325-018-0784-z. Epub 2018 Sep 12. PMID 30209750
- [Background] Cartwright TH, Parisi M, Espirito JL, Wilson TW, Pelletier C, Patel M, Babiker HM. Clinical Outcomes with First-Line Chemotherapy in a Large Retrospective Study of Patients with Metastatic Pancreatic Cancer Treated in a US Community Oncology Setting. Drugs Real World Outcomes. 2018 Sep;5(3):149-159. doi: 10.1007/s40801-018-0137-x. PMID 29946913
- [Background] Pelzer U, Wislocka L, Juhling A, Striefler J, Klein F, Roemmler-Zehrer J, Sinn M, Denecke T, Bahra M, Riess H. Safety and efficacy of Nab-paclitaxel plus gemcitabine in patients with advanced pancreatic cancer suffering from cholestatic hyperbilirubinaemia-A retrospective analysis. Eur J Cancer. 2018 Sep;100:85-93. doi: 10.1016/j.ejca.2018.06.001. Epub 2018 Jul 4. PMID 30014884
- [Background] Young R, Mainwaring P, Clingan P, Parnis FX, Asghari G, Beale P, Aly A, Botteman M, Romano A, Ferrara S, Margunato-Debay S, Harris M. nab-Paclitaxel plus gemcitabine in metastatic pancreatic adenocarcinoma: Australian subset analyses of the phase III MPACT trial. Asia Pac J Clin Oncol. 2018 Oct;14(5):e325-e331. doi: 10.1111/ajco.12999. Epub 2018 Jun 22. PMID 29932294
- [Background] Neumann CCM, von Horschelmann E, Reutzel-Selke A, Seidel E, Sauer IM, Pratschke J, Bahra M, Schmuck RB. Tumor-stromal cross-talk modulating the therapeutic response in pancreatic cancer. Hepatobiliary Pancreat Dis Int. 2018 Oct;17(5):461-472. doi: 10.1016/j.hbpd.2018.09.004. Epub 2018 Sep 7. PMID 30243879
- [Background] Veenstra VL, Damhofer H, Waasdorp C, van Rijssen LB, van de Vijver MJ, Dijk F, Wilmink HW, Besselink MG, Busch OR, Chang DK, Bailey PJ, Biankin AV, Kocher HM, Medema JP, Li JS, Jiang R, Pierce DW, van Laarhoven HWM, Bijlsma MF. ADAM12 is a circulating marker for stromal activation in pancreatic cancer and predicts response to chemotherapy. Oncogenesis. 2018 Nov 16;7(11):87. doi: 10.1038/s41389-018-0096-9. PMID 30442938
- [Background] Fernandez A, Salgado M, Garcia A, Buxo E, Vera R, Adeva J, Jimenez-Fonseca P, Quintero G, Llorca C, Canabate M, Lopez LJ, Munoz A, Ramirez P, Gonzalez P, Lopez C, Reboredo M, Gallardo E, Sanchez-Canovas M, Gallego J, Guillen C, Ruiz-Miravet N, Navarro-Perez V, De la Camara J, Ales-Diaz I, Pazo-Cid RA, Carmona-Bayonas A. Prognostic factors for survival with nab-paclitaxel plus gemcitabine in metastatic pancreatic cancer in real-life practice: the ANICE-PaC study. BMC Cancer. 2018 Nov 29;18(1):1185. doi: 10.1186/s12885-018-5101-3. PMID 30497432
- [Background] Hegewisch-Becker S, Aldaoud A, Wolf T, Krammer-Steiner B, Linde H, Scheiner-Sparna R, Hamm D, Janicke M, Marschner N; TPK-Group (Tumour Registry Pancreatic Cancer). Results from the prospective German TPK clinical cohort study: Treatment algorithms and survival of 1,174 patients with locally advanced, inoperable, or metastatic pancreatic ductal adenocarcinoma. Int J Cancer. 2019 Mar 1;144(5):981-990. doi: 10.1002/ijc.31751. Epub 2018 Oct 3. PMID 30006989
- [Background] Barnes JA, Ellis ML, Hwang S, Emarine J, Merwin P, Salinas GD, Musher BL. Identification of Educational Gaps Among Oncologists Who Manage Patients with Pancreatic Cancer. J Gastrointest Cancer. 2019 Mar;50(1):84-90. doi: 10.1007/s12029-017-0033-8. PMID 29177608
- [Background] Woo W, Carey ET, Choi M. Spotlight on liposomal irinotecan for metastatic pancreatic cancer: patient selection and perspectives. Onco Targets Ther. 2019 Feb 21;12:1455-1463. doi: 10.2147/OTT.S167590. eCollection 2019. PMID 30863113
- [Background] Sonbol MB, Ahn DH, Goldstein D, Okusaka T, Tabernero J, Macarulla T, Reni M, Li CP, O'Neil B, Van Cutsem E, Bekaii-Saab T. CanStem111P trial: a Phase III study of napabucasin plus nab-paclitaxel with gemcitabine. Future Oncol. 2019 Apr;15(12):1295-1302. doi: 10.2217/fon-2018-0903. Epub 2019 Feb 15. PMID 30768369